CLINICAL TRIAL: NCT03050840
Title: Gamification and Energetic Behavior Changes in Adolescent-Parent Dyads With Obesity
Brief Title: Gamification and Energetic Behavior Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-013613; 1UL1TR001878-01 (NIH)
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-monitoring (Other): Participants will wear a Fitbit, to self-monitor steps per day, and will report sugar sweetened beverage (SSB) consumption via text messaging. The Way to Health platform will record data.
  Interventions: Behavioral: Way to Health
- Self-monitoring plus gamification (Experimental): Participants will wear a Fitbit, to self-monitor steps per day, and will report sugar sweetened beverage consumption via text messaging. Participants will be awarded medals and points based on meeting step per day and SSB consumption goals The Way to Health platform will be used to record data.
  Interventions: Behavioral: Way to Health

INTERVENTIONS:
Behavioral: Way to Health — An online platform (Way to Health) will be used to test if self-monitoring plus gamification principles can increase steps per day and lower sugar sweetened beverage consumption per day, among obese children and adults, compared to self-monitoring alone.

SUMMARY:
Obesity [Body mass index (BMI kg/m2 ≥ 95th percentile)] affects 1 in 5 adolescents in the United States, with 13 million suffering from severe obesity (BMI ≥ 120% > 95th percentile or ≥ 35 mg/kg2). Adolescents are able to lose weight with behavioral changes in diet and physical activity, but change in these behaviors requires self-monitoring and support, and weight loss is not always successful.

Parent involvement and parent weight-loss can help their children to lose weight and successfully change their behavior. Guidance from pediatricians can also help to facilitate weight loss among obese adolescents. That said, treatment of obesity through behavior change within the time constraints of a Pediatric practice visit is limited by treatment adherence and clinic visit attendance. Therefore, finding cost-effective, timely, methods to keep adolescents with severe obesity engaged in therapy outside of standard practice is a critical need.

The effects of monetary incentives through games (gamification), and a comprehensive remote digital monitoring system on sleep, physical activity, and dietary intake, has been successful in adults, but has not been tested in adolescents with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Child Subjects age 10 - 16
* Obese as defined by body mass index (BMI)
* Computer access and data plan with text messaging
* SSB intake of 2 or more servings per day (1 serving=12oz)

Exclusion Criteria:

* Active substance abuse.
* Syndromic or secondary obesity.
* Any developmental disorder.
* Eating disorder (with the exception of binge eating disorder).
* Psychosis.
* Untreated depression.
* Use of medications (prescription or otherwise) known to effect body weight.
* Weight loss of more than 5% body weight in the past 3 months.
* History of bariatric surgery.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2018-01-27 (Actual)

PRIMARY OUTCOMES:
Difference in the total number of steps per day | 12 weeks
  Fitbit estimated steps per day will be compared between the two treatment groups at the end of the treatment period

SECONDARY OUTCOMES:
Difference in the total number of sugar sweetened beverages consumed per day | 12 weeks
  Self-reported sugar sweetened beverage consumption per day via automated text messaging and compared between the two groups at the end of the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Parks Prout, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No